CLINICAL TRIAL: NCT02841280
Title: Chlorthalidone in Chronic Kidney Disease
Acronym: CLICK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rajiv Agarwal, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1507540384
Record Dates: First submitted 2016-05-27; First posted 2016-07-22 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Renal Insufficiency, Chronic; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorthalidone (Experimental): Subjects with stage 4 chronic kidney disease (CKD) and poorly controlled hypertension confirmed by 24 hour ambulatory blood pressure monitoring will be randomized into two groups, one receiving placebo and one receiving a diuretic called chlorthalidone (12.5 mg at randomization). Doubling of the dose of the diuretic (up to 50 mg) or placebo will occur every 4 weeks if required by home blood pressure (BP) results.
  Interventions: Drug: Chlorthalidone
- Placebo (Placebo Comparator): Subjects with stage 4 CKD and poorly controlled hypertension confirmed by 24 hour ambulatory blood pressure monitoring will be randomized into two groups, one receiving placebo and one receiving a diuretic called chlorthalidone (12.5 mg at randomization). Doubling of the dose of the diuretic (up to 50 mg) or placebo will occur every 4 weeks if required by home BP results.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorthalidone — This is a forced-titration study and the study drug will be increased if goal BP is not achieved (dosage of chlorthalidone not to exceed 50 mg)
  Arms: Chlorthalidone
Drug: Placebo — This is a forced-titration study and placebo will be increased if goal BP is not achieved.
  Arms: Placebo

SUMMARY:
It is estimated that in the United States there are approximately 8 million individuals who have moderate to severe chronic kidney disease (CKD). Among them hypertension is common and is often poorly controlled due to an expanded volume state; diuretics are frequently prescribed. Loop diuretics are potent and effective in lowering blood pressure (BP) but their use is associated with acute kidney injury. Thiazide diuretics, on the other hand, are less potent, their use may be associated with less acute kidney injury, but as yet there are no firm data to support that thiazide diuretic therapy can improve BP among subjects with advanced CKD. The investigators found 13 studies on the use of thiazide diuretics in advanced CKD either alone or in combination with loop diuretics and concluded that thiazides may be useful. Thiazides cause a negative Na balance, increase Na excretion by 10-15% and weight loss by 1-2 kg in observational studies. Observational data show that thiazides lead to an improvement in seated clinic BP of about 10-15 mmHg systolic and 5-10 mmHg diastolic whereas randomized trials show about a 15 mmHg reduction in mean BP. Randomized trials had only between 7 and 23 subjects each; accordingly, larger studies are needed to evaluate their safety and efficacy in moderate to advanced CKD.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blind, randomized controlled trial of chlorthalidone (CTD) in patients with CKD and poorly controlled hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years.
2. Calculated glomerular filtration rate (GFR) by 4-component Modification of Diet in Renal Disease (MDRD) formula < 30 ml/min/1.73m2 but ≥15 mL/min/1.73m2. The hospital laboratory uses isotope dilution mass spectrometry (IDMS) calibrated creatinine and the appropriate formula is used to estimate GFR.
3. Hypertension. This is defined as BP of either ≥130 systolic or ≥80 mmHg by 24-hour ambulatory BP monitoring.
4. Treatment with antihypertensive drugs: This would require the use of at least one antihypertensive drug. One of the drugs should be either an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB). If these are contraindicated then use of a beta-blocker is required prior to randomization.

Exclusion Criteria:

1. Use of thiazide or thiazide-like drugs in the previous 12 weeks.
2. Use of furosemide in a dose >200 mg/d.
3. BP of either ≥160 systolic or ≥100 mmHg by 24-hour ambulatory BP monitoring.
4. Expected to receive renal replacement therapy within the next 3 months.
5. Myocardial infarction, heart failure hospitalization, or stroke ≤3 months prior to randomization.
6. Pregnant or breastfeeding women or women who are planning to become pregnant or those not using a reliable form of contraception (oral contraceptives. condoms and diaphragms will be considered reliable).
7. Known hypersensitivity to thiazide or sulfa drugs.
8. Organ transplant recipient or therapy with immunosuppressive agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Division of Nephrology, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Agarwal R, Sinha AD, Cramer AE, Balmes-Fenwick M, Dickinson JH, Ouyang F, Tu W. Chlorthalidone for Hypertension in Advanced Chronic Kidney Disease. N Engl J Med. 2021 Dec 30;385(27):2507-2519. doi: 10.1056/NEJMoa2110730. Epub 2021 Nov 5. PMID 34739197
- [Derived] Agarwal R, Cramer AE, Balmes-Fenwick M, Sinha AD, Ouyang F, Tu W. Design and Baseline Characteristics of the Chlorthalidone in Chronic Kidney Disease (CLICK) Trial. Am J Nephrol. 2020;51(7):542-552. doi: 10.1159/000508700. Epub 2020 Jul 14. PMID 32663820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by screening for potential participants for eligibility at 3 medical centers between June 29, 2016 and January 7, 2021. The first participant consented on July 14, 2016, and the last participant was randomized on January 20, 2021.
Pre-assignment Details: Of the 403 consented patients, 160 met inclusion criteria and were randomized to treatment. Thus, 160 are considered enrolled for the purposes of this report.
Groups:
- Chlorthalidone: Subjects with stage 4 chronic kidney disease (CKD) and poorly controlled hypertension confirmed by 24 hour ambulatory blood pressure monitoring will be randomized into two groups, one receiving placebo and one receiving a diuretic called chlorthalidone (12.5 mg at randomization). Doubling of the dose of the diuretic (up to 50 mg) or placebo will occur every 4 weeks if required by home blood pressure (BP) results.
  Chlorthalidone: This is a forced-titration study and the study drug or placebo will be increased if goal BP is not achieved (dosage of chlorthalidone not to exceed 50 mg)
- Placebo: Subjects with stage 4 CKD and poorly controlled hypertension confirmed by 24 hour ambulatory blood pressure monitoring will be randomized into two groups, one receiving placebo and one receiving a diuretic called chlorthalidone (12.5 mg at randomization). Doubling of the dose of the diuretic (up to 50 mg) or placebo will occur every 4 weeks if required by home BP results.
  Placebo: This is a forced-titration study and the study drug or placebo will be increased if goal BP is not achieved (dosage of chlorthalidone not to exceed 50 mg)
Period: Overall Study
Arm/Group | Chlorthalidone | Placebo
Started | 81 | 79
Completed | 67 | 73
Not Completed | 14 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Stop Point: BP above threshold | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorthalidone | Placebo | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 47 | 46 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (10.8) | 66.7 (10.8) | 66.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 62 | 62 | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnic Group: White | 46 | 47 | 93
  Race or Ethnic Group: Black | 32 | 32 | 64
  Race or Ethnic Group: Asian | 2 | 0 | 2
  Race or Ethnic Group: Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 81 | 79 | 160
Medical History of Diabetes Mellitus [Count of Participants; unit: Participants] | 60 | 61 | 121
Cause of Chronic Kidney Disease [Count of Participants; unit: Participants]
  Diabetes | 42 | 42 | 84
  Hypertension | 26 | 26 | 52
  Glomerulonephritis | 3 | 5 | 8
  Obstructive Uropathy | 3 | 2 | 5
  Polycystic Kidney Disease | 1 | 1 | 2
  Other | 6 | 3 | 9
Current Smoking [Count of Participants; unit: Participants] | 21 | 19 | 40
Height [Mean (Standard Deviation); unit: cm] | 171.7 (11.3) | 173.0 (8.6) | 172.3 (10.1)
Weight [Mean (Standard Deviation); unit: kg] | 97.4 (23.6) | 95.8 (23.5) | 96.6 (23.6)
Body-Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.0 (7.0) | 32.0 (7.4) | 32.5 (7.2)
Hip Circumference [Mean (Standard Deviation); unit: cm] | 115.9 (14.9) | 114.6 (15.0) | 115.3 (14.9)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 115.3 (17.0) | 115.4 (16.6) | 115.3 (16.8)
Waist-to-Hip Ratio [Mean (Standard Deviation); unit: ratio] | 1.011 (0.078) | 0.998 (0.074) | 1.005 (0.076)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 141.2 (15.1) | 138.7 (16.0) | 140.0 (15.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 69.2 (12.3) | 67.9 (13.9) | 68.6 (13.1)
Pulse Rate [Mean (Standard Deviation); unit: beats/min] | 66.5 (11.7) | 64.3 (11.1) | 65.4 (11.4)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: ml/min/1.73 m^2] | 23.5 (4.2) | 22.8 (4.2) | 23.2 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Weeks in Systolic Ambulatory Blood Pressure in the Chlorthalidone Group Compared to Placebo.
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Chlorthalidone | Placebo
Number analyzed (Participants) | 81 | 79
mm Hg | -11.0 [-13.9 to -8.1] | -0.5 [-3.5 to 2.5]

2. Secondary Outcome: Changes in Albuminuria From Baseline at Each 4 Week Visit in the Log Transformed Albumin/Creatinine Ratio in the Chlorthalidone Group Compared to Placebo
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change in UACR
Arm/Group | Chlorthalidone | Placebo
Number analyzed (Participants) | 81 | 79
percentage of change in UACR
  Percent change in albuminuria 4 weeks from baseline in UACR | -41 [-49 to -30] | -7 [-20 to 9]
  Percent change in albuminuria 8 weeks from baseline in UACR | -45 [-53 to -35] | -3 [-17 to 13]
  Percent change in albuminuria 12 weeks from baseline in UACR | -52 [-59 to -43] | -4 [-18 to 12]

3. Secondary Outcome: Change From Baseline at Each 4 Week Visit in Log of Aldosterone and Log of Renin in the Chlorthalidone Group Compared to Placebo. No Adjustments Will be Made for Multiple Comparisons.
Time Frame: Baseline to 12 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Chlorthalidone | Placebo
Number analyzed (Participants) | 81 | 79
percentage of change
  Percent change 4 weeks from baseline in aldosterone | 57 [34 to 84] | 16 [-1 to 36]
  Percent change 8 weeks from baseline in aldosterone | 65 [40 to 95] | 12 [-4 to 32]
  Percent change 12 weeks from baseline in aldosterone | 52 [28 to 79] | 8 [-8 to 27]
  Percent change 4 weeks from baseline in renin | 57 [45 to 70] | 14 [5 to 23]
  Percent change 8 weeks from baseline in renin | 67 [54 to 81] | 5 [-3 to 14]
  Percent change 12 weeks from baseline in renin | 64 [50 to 78] | 15 [6 to 25]

4. Secondary Outcome: Change From Baseline at Each 4 Week Visit in Log of N-terminal Pro B-type Natriuretic Peptide (NTproBNP) in the Chlorthalidone Group Compared to Placebo. No Adjustments Will be Made for Multiple Comparisons.
Time Frame: Baseline to 12 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of change in NTproBNP
Arm/Group | Chlorthalidone | Placebo
Number analyzed (Participants) | 81 | 79
percentage of change in NTproBNP
  Percent change from 4 weeks from baseline in NTproBNP | -25 [-36 to -14] | -14 [-26 to 0]
  Percent change from 8 weeks from baseline in NTproBNP | -32 [-42 to -21] | 5 [-9 to 22]
  Percent change from 12 weeks from baseline in NTproBNP | -30 [-39 to -19] | -11 [-23 to 2]

5. Secondary Outcome: Change From Baseline at Each 4 Week Visit in Body Volume in the Chlorthalidone Group Compared to Placebo. No Adjustments Will be Made for Multiple Comparisons.
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Chlorthalidone | Placebo
Number analyzed (Participants) | 81 | 79
Liters
  Change in body volume 4 weeks from baseline | -1.1 [-1.7 to -0.6] | 0.2 [-0.3 to 0.7]
  Change in body volume 8 weeks from baseline | -1.7 [-2.2 to -1.1] | 0.3 [-0.2 to 0.8]
  Change in body volume 12 weeks from baseline | -2 [-2.6 to -1.5] | 0.3 [-0.3 to 0.8]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the period from the time of randomization to the discontinuation of the regimen (12 weeks).
Arm/Group | Chlorthalidone | Placebo
All-Cause Mortality (participants affected / at risk) | 1/81 | 0/79
Serious Adverse Events (participants affected / at risk) | 8/81 | 11/79
Other Adverse Events (participants affected / at risk) | 74/81 | 68/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorthalidone (N=81) | Placebo (N=79)
Infection (Infections and infestations) | 2 (3) | 1 (1)
Cardiovascular Event (Cardiac disorders) | 3 (3) | 5 (7)
Renal Event (Renal and urinary disorders) | 1 (1) | 1 (1)
Event of Interest (General disorders) | 3 (4) | 0 (0) — Event of Interest included orthostatic hypotension, acute kidney injury, hyperglycemia, and hypokalemia
Other (General disorders) | 3 (3) | 5 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorthalidone (N=81) | Placebo (N=79)
Infection (Infections and infestations) | 6 (6) | 10 (10)
Cardiovascular Event (Cardiac disorders) | 2 (2) | 3 (3)
Other (General disorders) | 42 (57) | 39 (64)
Hypokalemia (Renal and urinary disorders) | 8 (10) | 0 (0)
Hypomagnesemia (Renal and urinary disorders) | 19 (35) | 13 (26)
Hyponatremia (Renal and urinary disorders) | 9 (12) | 6 (6)
Hypocalcemia (Renal and urinary disorders) | 1 (1) | 1 (3)
Hypercalcemia (Renal and urinary disorders) | 2 (3) | 2 (3)
Hyperglycemia (Renal and urinary disorders) | 13 (18) | 4 (5)
Hyperuricemia (Renal and urinary disorders) | 16 (32) | 7 (9)
Hyperkalemia (Renal and urinary disorders) | 5 (5) | 7 (8)
Hypernatremia (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Gout (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Syncope (Cardiac disorders) | 2 (2) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 8 (12) | 5 (8) — Orthostatic hypotension was defined as a decrease in the standing systolic blood pressure greater than 20 mm Hg, accompanied by a feeling of dizziness or light-headedness.
Dizziness (Cardiac disorders) | 20 (33) | 13 (24) — Dizziness was recorded when the patient felt dizzy when standing from a seated position but did not have a decrease in the systolic blood pressure greater than 20 mm Hg.
Asymptomatic Orthostatic Hypotension (Vascular disorders) | 21 (39) | 18 (33) — Asymptomatic orthostatic hypotension was defined as a decrease in the standing systolic blood pressure greater than 20 mm Hg that was not accompanied by a feeling of dizziness or light-headedness.
Acute Kidney Injury (Renal and urinary disorders) | 33 (61) | 10 (12)

LIMITATIONS AND CAVEATS:
The trial was relatively small and had an underrepresentation of women (36 of 160 patients [22%] were women). In addition, very few patients were Asian or Hispanic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT02841280/Prot_SAP_000.pdf